CLINICAL TRIAL: NCT05996094
Title: Adherence and Pharmacokinetics Measures in People Living With HIV Receiving Tenofovir Disoproxil Fumarate-based Regimens in Indonesia
Brief Title: Antiretroviral Adherence and Drug-level Monitoring
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Zamrotul Izzah (Other)
Collaborators: Universitas Airlangga (Other)
Responsible Party: Sponsor-Investigator, Zamrotul Izzah, Principal Investigator, University of Groningen
Organization: University of Groningen (Other)
Other Study IDs: 3578141P111242020012800013
Record Dates: First submitted 2023-07-21; First posted 2023-08-16 (Actual); Last update posted 2023-08-21 (Actual); Status verified 2023-08

CONDITIONS: HIV Infections; AIDS; Antiretroviral Therapy, Highly Active; Adherence, Medication; Drug-level Monitoring
Keywords: Adherence; Adult; Pharmacokinetics; Tenofovir; Viral Load
MeSH Terms: conditions — HIV Infections; Acquired Immunodeficiency Syndrome; Medication Adherence

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This observational study aims to investigate medication adherence and drug-level monitoring of antiretroviral agents in a cohort of people living with HIV in Indonesia. The study is conducted in outpatients receiving tenofovir-based regimens in a university medical centre.

DETAILED DESCRIPTION:
Optimal adherence is critical to achieve and sustain viral suppression. Currently, there is no gold standard measure of antiretroviral adherence and exposure in clinical practice. Recent studies have evaluated the use of emerging biological matrices such as dried blood spots, urine, and saliva as means of objective adherence measures. For drug-level monitoring, tenofovir is selected as a drug of interest and thus only people receiving tenofovir disoproxil fumarate-based regimens will be monitored. Some studies have reported that higher plasma trough concentrations of tenofovir were associated with renal toxicity. Therefore, this project aims to measure level of adherence and tenofovir concentrations in plasma and emerging matrices among people living with HIV in Indonesia. Primary outcome is adherence to ART that will be measured using multi methods, including self-report questionnaire, pill counting, electronic monitoring, and drug-level testing. Secondary outcomes include tenofovir concentrations in plasma, urine, saliva, and dried blood spots and clinical outcomes (viral load and CD4 count). Assays for measuring tenofovir concentrations will be developed using high-performance liquid chromatography-tandem mass spectrometry. Concentrations derived from dried blood spots, saliva, and urine will be compared to plasma concentrations. Pharmacokinetic models will be used to interpret drug-level monitoring. The association of adherence measures as well as drug concentrations and clinical outcomes will be examined.

ELIGIBILITY:
Inclusion Criteria:

* Adults with HIV who have been receiving antiretroviral therapy containing tenofovir-based regimens for at least six months

Exclusion Criteria:

* Pregnant and breastfeeding women, people with kidney failure, undergoing hemodialysis or peritoneal dialysis, uncontrolled diabetes, uncontrolled hypertension, and hypersensitivity to tenofovir

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All people living with HIV receiving antiretroviral therapy who regularly visit the HIV clinic at a university medical centre in Surabaya, Indonesia, during study period.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2020-10-16 (Actual); Primary Completion 2023-12-31 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
Adherence to antiretroviral therapy | Baseline and 6 months
  Adherence to antiretroviral therapy (ART) will be assessed using a validated Bahasa Indonesia version of self-reported adherence questionnaire. The questionnaire will recall ART use in the past week, past month, and past three months. The percentages of adherence will be calculated by the formula: (total number of dosage units prescribed - total number of times reported) / (total number of dosage units prescribed) × 100. The adherence scales range from 0 to 100% with higher scales denote higher adherence. Being highly adherent to ART is defined by having an adherence higher than 80%.

SECONDARY OUTCOMES:
Tenofovir concentrations | Baseline (pre-dose, 1, and 4 h post-dose) and 6 months (random 3 - 16 h post-dose)
  Concentrations of tenofovir in plasma, saliva, urine, and dried blood spots
Viral load | Baseline and 6 months
  The viral load test will measure the number of HIV copies in plasma (in copies/ml).
CD4 cell count | Baseline and 6 months
  The cluster of differentiation 4 (CD4) cell count test will quantify CD4 cells in plasma (in cells/mm^3).

CONTACTS AND LOCATIONS:
Overall Officials: Zamrotul Izzah, Principal Investigator — Universitas Airlangga
Locations (1):
- Universitas Airlangga Hospital, Surabaya, East Java, Indonesia

IPD SHARING:
Plan to Share IPD: No
De-identified data will be available for analysing and reporting purposes and for other parties upon formal request to the principal investigators.